CLINICAL TRIAL: NCT03661788
Title: Network Connectivity and Inhibitory Control Under Atomoxetin Challenge- A Pharmacological 'Resting State' and 'Inhibiton Task' Study in Patients With ADHD
Acronym: CAIAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 11-185 CAIAC; 2013-002386-18 (EudraCT Number)
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: ADHD
Keywords: Atomoxetin; fMRT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- First placebo, than atomoxetin (Experimental): Patients receive a placebo in the first of the two 14-day treatment intervals and atomoxetin in the second 14-day treatment intervals. Between the treatment intervals there is a wash-out phase of two weeks. The order of treatment is randomized.
  Interventions: Drug: Atomoxetine; Drug: Placebos
- First atomoxetin, than placebo (Experimental): Patients receive atomoxetin in the first of the two 14-day treatment intervals and a placebo in the second 14-day treatment interval. Between the treatment intervals there is a wash-out phase of two weeks. The order of treatment is randomized.
  Interventions: Drug: Atomoxetine; Drug: Placebos

INTERVENTIONS:
Drug: Atomoxetine — 14-day treatment interval: first week 40 mg atomoxetine (one pill), second week 80mg atomoxetine (two pills)
  Other Names: Strattera
Drug: Placebos — 14-day treatment interval: first week one placebo pill, second week two placebo pills

SUMMARY:
Attention deficit /hyperactivity disorder (ADHD) is a disorder which manifests in childhood but often persists through adulthood. The most prominent symptoms in adults are inattention, emotional instability, disorganized behavior, impulsivity and restlessness, which cause several restrictions in different areas of life. It is suggested that those symptoms can be attributed to a general deficit in inhibitory control. This hypothesis is supported by several studies revealing that patients with ADHD show poor performance completing inhibitory control tasks.

Furthermore, studies showed that a unique administration of atomoxetin (ATX) significantly improves inhibitory control in patients with ADHD as well as in healthy participtants. In contrast to other medication authorized for the treatment of patients with ADHD, does ATX has no risk for potential addiction. Due its indirect mode of action, ATX has a delayed effect occurence taking up to 2 weeks. However, this apects was unconsidered in those studies.

Although we directly often associate failures in cognitive control with disruptions at prefrontal areas of the brain, there exists a specific brain network which is called the default mode network (DMN), which is suggested to be at least partly responsibe for the ADHD symptomatic.

The following study is interested in which way a 2- week intake of ATX affects the DMN and surrounding networks in their connectivity during a inhibitory control task and during rest in patients with ADHD vs controls.

ELIGIBILITY:
Inclusion Criteria:

* Male Age 18-45 years Diagnosis of ADHD (patients) or no axis I disorder (controls) according the DSM IV No substance abuse/ dependency Understanding of the study information and declaration of agreement Ability to read, understand and speak German No severe medical disorders No risk for suicide

Exclusion Criteria:

* Drug dependence or the a positive drug screening Other Severe physical disorders Current pharmacological therapy because of another psychiatric disorder Risk for seizure or cardiac problems Impaired liver and renal function Significant deviations in regard to clinical chemistry, haematology or EKG Relationship of dependency with the sponsor or the investigator Unable to keep to the study protocol Known Intolerance of the study medication fMRI scanner incompatibility

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12-06 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
FMRT resting state connecitivty of the default mode network | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded into the data pool of the Deutsches Netzwerk zu psychischen Erkrankungen.